CLINICAL TRIAL: NCT05412160
Title: Improving Quality of Life and Daily Life Activities With Bioarginine in Patients With COPD: a Multicenter, Randomized, Controlled, Proof of Concept Study
Brief Title: Improving Quality of Life and Daily Life Activities With Bioarginine in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOCOPD2022
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: COPD; Dyspnea; Argininemia
Keywords: COPD; Arginine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Hyperargininemia | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A - BioArginine receivers (Experimental): Patients will be randomized to receive BioArginine C™ twice daily on top of usual chronic inhaled therapy
  Interventions: Drug: Arginine
- ARM B - placebo receivers (Placebo Comparator): Patients will be randomized to receive placebo twice daily on top of usual chronic inhaled therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arginine — During the first assessment the patients will be randomized to receive BioArginine C™ twice daily on top of chronic inhaled therapy or to continue their chronic Inhaled therapy plus placebo for 6 weeks. The main purpose is to compare changes in CRQ from baseline and after 6 weeks in the interventional arm compared with the control group in order to evaluate whether in symptomatic patients with COPD, daily bioarginine on top of chronic inhaled therapy can improve respiratory symptoms and dyspnea. The secondary objective of the study is to determine whether there is any correlation between improvement in respiratory symptoms and distance walked at the 6MWT and lung function parameters.
  Arms: ARM A - BioArginine receivers
Drug: Placebo — During the first assessment the patients will be randomized to receive BioArginine C™ twice daily on top of chronic inhaled therapy or to continue their chronic Inhaled therapy plus placebo for 6 weeks. The main purpose is to compare changes in CRQ from baseline and after 6 weeks in the interventional arm compared with the control group in order to evaluate whether in symptomatic patients with COPD, daily bioarginine on top of chronic inhaled therapy can improve respiratory symptoms and dyspnea. The secondary objective of the study is to determine whether there is any correlation between improvement in respiratory symptoms and distance walked at the 6MWT and lung function parameters.
  Arms: ARM B - placebo receivers

SUMMARY:
Different studies have suggested that COPD is associated with elevated alveolar NO and increased expression of NOS2 in alveolar walls, small airway epithelium and vascular smooth muscle. Furthermore, arginase activity in COPD is shown to correlate inversely with total NO metabolite in sputum and with pre- and post- bronchodilator FEV1; at the same time ADMA levels in serum is shown to be correlated with airway resistance and ADMA in COPD airways was documented to be able to shift the L-arginine metabolism towards the arginase pathway. As demonstrated in a guinea pig model, the arginase inhibition can shift the L-ornitine: L-citrulline ratio towards L-citrulline, preventing neutrophilia, mucus hypersecretion and collagen synthesis. Thus, increasing substrate availability for NOS by arginase inhibition or supplementation of L-arginine or L-citrulline or a combination thereof, may represent a window of opportunity in patients with COPD.

The present study was constructed in order to investigate as a primary objective whether in symptomatic patients with COPD, daily bioarginine on top of chronic inhaled therapy can improve patients' respiratory symptoms and dyspnea during daily life activities. The secondary objective of the study is to determine whether there is any correlation between improvement in respiratory symptoms and distance walked at the 6MWT and lung function parameters. In order to do so, the investigators designed a multi center, interventional, prospective, randomized, controlled vs placebo, proof of concept study: COPD patients will be randomized to receive BioArginine twice daily on top of chronic inhaled therapy or to continue their chronic Inhaled therapy plus placebo for 6 weeks. In order to evaluate the impact on respiratory symptoms and dyspnea the CRQ (Chronic Respiratory disease Questionnaire) and the LCADL (London Chest Activities of daily Living) Scale, as well as the 6MWT, will be used.

ELIGIBILITY:
Inclusion Criteria:

* > 40 years old
* Smoke history >10 pack years (PYs)
* Forced expiratory volume (FEV1 70-40% predicted)
* COPD Assessment Test score >= 10
* Stable Inhaled therapy in the three months prior to study enrollment

Exclusion Criteria:

* Exacerbations in the three months prior to study enrolment
* Dementia and inability to perform study test bundles
* Interstitial lung disease
* History of asthma
* Patients unable to perform a 6MWT or necessitating a walker to ambulate
* Long term oxygen therapy (excluding patients on nocturnal O2 therapy)
* Patients enrolled In pulmonary rehabilitation programs during the study or that have completed a pulmonary rehabilitation program in the 6 months before study enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
To compare changes in CRQ from baseline and after 6 weeks in the interventional arm compared with the control group | 6 weeks
  Patients will undergo the assesment of the Chronic Respitatory Qestionnaire at the time of study erollment and after 6 weeks of treatment with bioarginine or placebo.
  The questionnaire contains 20 questions which can be divided into four domains:
  * Dyspnoea (5 questions), The dyspnoea domain is "individualised" which means that it is made up of five activities chosen by a patient to cause the greatest shortness of breath. The patient then rates the dyspnoea on these self-selected activities during subsequent administrations of the CRQ.
  * Fatigue (4 questions),
  * Emotional functioning (7 questions),
  * Mastery (4 questions).
  * Answers can be scored on a seven point scale ranging from 1 which indicates maximum impairment to 7 which indicates no impairment. The results are expressed as the mean score for each domain and the mean overall score.
  * The minimally important difference was found to be an improvement (or deterioration) of 0.5

SECONDARY OUTCOMES:
To compare changes in LCADL from baseline and after 6 weeks in the interventional arm compared with the control group | 6 weeks
  Patients will undergo the assesment of the London Chest Activities of Daily Living at the time of study erollment and after 6 weeks of treatment with bioarginine or placebo.
  The LCADL scale is a 15-item tool that measures the effect of dyspnea on routine daily activities. The LCADL provides a total score from 0 to 75 points with higher scores indicating greater limitations. Domain scores include personal care (0-20), domestic activities (0-30), physical activity (0-10), and leisure (0-15). The minimal detectable change (MDC) for the total score is 3.88 or approximately 4 points, 0.89 for personal care, 2.60 for domestic activities, 0.44 for physical activities, and 0.58 for leisure.
  The minimal detectable change (MDC) for the total score is 3.88 or approximately 4 points, 0.89 for personal care, 2.60 for domestic activities, 0.44 for physical activities, and 0.58 for leisure.
To compare changes in the distance covered during the 6MWT from baseline and after 6 weeks in the interventional arm compared with the control group | 6 weeks
  Patiens will undergo the Six Minutes Walking Test at study enrolment and after 6 weeks of treatment with bioarginine or placebo.
  The 6MWT will be conducted in room air conditions, in a corridor of 30 meters of lenght while the patients has being monitored with a pulsoxymeter that will register the peripheral oxygen saturation and heart right during the test. At the beginning and at the end of the test, Borg Dyspnea Scale (0-10 points), blood pressure and vitals will be registered. The patient will be asked to walk with a sutained pace for six minutes and the distance covered will be recorded. The mMCID of the 6MWT has been definied of 40 meter.
To compare changes in the dyspnea domain of the CRQ from baseline and after 6 weeks in the interventional arm compared with the control group | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jaeschke R, Singer J, Guyatt GH. Measurement of health status. Ascertaining the minimal clinically important difference. Control Clin Trials. 1989 Dec;10(4):407-15. doi: 10.1016/0197-2456(89)90005-6. PMID 2691207
- [Background] Bisca GW, Proenca M, Salomao A, Hernandes NA, Pitta F. Minimal detectable change of the London chest activity of daily living scale in patients with COPD. J Cardiopulm Rehabil Prev. 2014 May-Jun;34(3):213-6. doi: 10.1097/HCR.0000000000000047. PMID 24531202
- [Background] Garrod R, Bestall JC, Paul EA, Wedzicha JA, Jones PW. Development and validation of a standardized measure of activity of daily living in patients with severe COPD: the London Chest Activity of Daily Living scale (LCADL). Respir Med. 2000 Jun;94(6):589-96. doi: 10.1053/rmed.2000.0786. PMID 10921765
- See also: CRQ questionnaire — https://qol.thoracic.org/sections/instruments/ae/pages/crq.html